CLINICAL TRIAL: NCT00116558
Title: Early Treatment of Amyotrophic Lateral Sclerosis With Nutrition and Non-Invasive Positive Pressure Ventilation
Brief Title: Early Treatment of Amyotrophic Lateral Sclerosis (ALS) With Nutrition and Non-Invasive Positive Pressure Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edward Kasaraskis (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Edward Kasaraskis, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R01NS045087 (NIH); R01NS045087 (NIH)
Record Dates: First submitted 2005-06-29; First posted 2005-06-30 (Estimated); Results first posted 2019-07-31 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: amyotrophic lateral sclerosis; ALS; Lou Gehrig's disease; nutrition; NIPPV; non-invasive positive pressure ventilation; percutaneous endoscopic gastrostomy; PEG
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Early NIPPV Intervention (Experimental): Participants with >80% predicted forced vital capacity (FVC).
  Interventions: Device: Early NIPPV
- Standard of Care NIPPV (Active Comparator): Participants with 50-74% predicted forced vital capacity (FVC).
  Interventions: Device: Standard NIPPV
- Standard of Care NIPPV and Nutritional Monitoring (Active Comparator): Participants with 50-95% forced vital capacity (FVC), and normal or impaired amyotrophic lateral sclerosis functional rating scale (ALSFRS) scores. Participants in this group will receive standard of care NIPPV therapy but will also undergo detailed analysis of nutritional status.
  Interventions: Device: Standard NIPPV

INTERVENTIONS:
Device: Early NIPPV — Early intervention with non-invasive positive pressure ventilation (NIPPV) at 80% forced vital capacity (FVC).
  Other Names: BiPAP (Bilevel Positive Airway Pressure)
  Arms: Early NIPPV Intervention
Device: Standard NIPPV — Standard of care non-invasive positive pressure ventilation (NIPPV) at 50% forced vital capacity (FVC).
  Other Names: BiPAP (Bilevel Positive Airway Pressure)
  Arms: Standard of Care NIPPV; Standard of Care NIPPV and Nutritional Monitoring

SUMMARY:
The purposes of the study are to determine the energy balance and evaluate the nutritional status of patients with ALS, and to investigate the use of NIPPV as respiratory support to treat patients with ALS.

DETAILED DESCRIPTION:
Studies to date indicate that percutaneous endoscopic gastrostomy (PEG)-insertion of a feeding tube in the stomach-and non-invasive positive pressure ventilation (NIPPV)-mechanically assisted or generated breaths delivered through a tightly fitting nasal or facial mask-improve survival in amyotrophic lateral sclerosis (ALS), even when introduced late in the disease.

Dr. Kasarskis and his research team believe early intervention with these treatments may improve patients outcome even further. However, many issues regarding the early use of these treatments prevent the design of a phase III clinical trial to test this hypothesis. Common to both NIPPV and nutrition is a lack of a reliable indicator of early respiratory or nutritional insufficiency. With respect to nutrition, reliable and cost effective methods are needed to determine a patient's energy (i.e. caloric) requirements at different stages of the illness to establish a basis for recommending PEG on the adequacy of energy intake. For NIPPV, factors that influence acceptance and tolerability of this therapy, and measurements of early respiratory dysfunction need to be identified.

The purposes of this trial are to develop and validate strategies to improve tolerability of NIPPV, identify factors that influence acceptance of NIPPV, and evaluate measures of early respiratory failure, other than percentage of forced vital capacity (FVC). Researchers will also develop and validate methods to determine energy balance in and evaluate the nutritional status of patients with ALS that will be applicable to a multi-center phase III study of nutrition and NIPPV.

The study will be conducted at 11 other sites across the country. Some study sites will focus on the nutritional aspects of the trial while the other sites will focus on NIPPV treatment. A total of 220 patients will be studied over 2 years.

Enrollment will end on June 30, 2007. The last patient was followed clinically until June 30, 2008. The study remained open for sample analysis, data analysis, and assessment of vital status until the completion of funding on November 30, 2009.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent.
* If women of childbearing age, must be non-lactating and surgically sterile or using an effective method of birth control (double-barrier or oral contraception) and have a negative pregnancy test.
* Minorities: All races and ethnic backgrounds.
* Disease inclusion: Clinically possible/definite/probable, or laboratory supported probable, sporadic or familial ALS according to the revised Escorial criteria.
* Onset of progressive weakness within 60 months prior to study.
* Willing to return for visits as scheduled and adhere to protocol requirements.

FVC Criteria

* NIPPV Arm: Best-sitting FVC between 50% and 95% of predicted normal.
* Nutrition Arm: Best-sitting FVC >50% of predicted normal.

Exclusion Criteria:

* Untreated or unstable hyper or hypothyroidism, untreated or unstable asthma, unstable angina, advanced liver or renal disease, advanced cancer, untreated diabetes or chronic obstructive pulmonary disease (COPD).
* Diagnosis of other motor neuron or other neurological disorder that mimics ALS.
* Diagnosis of other neurodegenerative disease (i.e., Parkinson's disease, Alzheimer's disease, etc.)
* Inflammatory bowel disease or malabsorption syndrome.
* Use of NIPPV, mechanical ventilation, or tracheostomy at the time of consent.
* Inability to adhere to study visit schedule or lack of reliable caretaker if participant requires one.
* Pregnant or lactating woman.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2004-08-01 (Actual); Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Kasarskis, MD, PhD, Principal Investigator — University of Kentucky
Locations (12):
- United States (12):
  - University of Colorado, Denver, Colorado
  - University of Miami, Miami, Florida
  - University of Kentucky, Lexington, Kentucky
  - Henry Ford Hospital, Detroit, Michigan
  - Beth Israel, New York, New York
  - Columbia University, New York, New York
  - SUNY, Syracuse, New York
  - Pennsylvania State University, Hershey, Pennsylvania
  - Drexel University, Philadelphia, Pennsylvania
  - University of Texas-San Antonio, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Vermont, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kasarskis EJ, Mendiondo MS, Matthews DE, Mitsumoto H, Tandan R, Simmons Z, Bromberg MB, Kryscio RJ; ALS Nutrition/NIPPV Study Group. Estimating daily energy expenditure in individuals with amyotrophic lateral sclerosis. Am J Clin Nutr. 2014 Apr;99(4):792-803. doi: 10.3945/ajcn.113.069997. Epub 2014 Feb 12. PMID 24522445
- [Background] Scagnelli CN, Howard DB, Bromberg MB, Kasarskis EJ, Matthews DE, Mitsumoto HM, Simmons Z, Tandan R; ALS Nutrition-NIPPV Study Group. Hydration measured by doubly labeled water in ALS and its effects on survival. Amyotroph Lateral Scler Frontotemporal Degener. 2018 May;19(3-4):220-231. doi: 10.1080/21678421.2017.1413117. Epub 2017 Dec 15. PMID 29243507
- [Result] Kasarskis EJ, Mendiondo MS, Wells S, Malguizo MS, Thompson M, Healey M, Kryscio RJ; ALS Nutrition/NIPPV Study Group. The ALS Nutrition/NIPPV Study: design, feasibility, and initial results. Amyotroph Lateral Scler. 2011 Jan;12(1):17-25. doi: 10.3109/17482968.2010.515225. PMID 21271789

RESULTS

PARTICIPANT FLOW:
Groups:
- Early NIPPV: Participants with >80% predicted forced vital capacity (FVC).
Period: Overall Study
Arm/Group | Standard of Care NIPPV and Nutritional Monitoring | Standard of Care NIPPV | Early NIPPV
Started | 80 | 26 | 47
Completed | 49 | 11 | 14
Not Completed | 31 | 15 | 33
Not completed — Death | 11 | 5 | 3
Not completed — Withdrawal by Subject | 17 | 3 | 12
Not completed — disease progression | 3 | 7 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care NIPPV and Nutritional Monitoring | Standard of Care NIPPV | Early NIPPV Intervention | Total
Number analyzed (Participants) | 80 | 26 | 47 | 153
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (11.7) | 60.8 (11.4) | 56.2 (11.2) | 58.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 10 | 17 | 55
  Male | 52 | 16 | 30 | 98
Region of Enrollment [Number; unit: participants]
  United States | 80 | 26 | 47 | 153

OUTCOME MEASURES:

1. Primary Outcome: Acceptance Rate of Early Non-invasive Positive Pressure Ventilation (NIPPV) Treatment.
Description: Percentage of patients attempting to use NIPPV therapy within six weeks of initial offer.
Time Frame: 6 weeks
Population: Data were not obtained from the "Standard of Care NIPPV and Nutritional Monitoring" arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care NIPPV and Nutritional Monitoring | Standard of Care NIPPV | Early NIPPV Intervention
Number analyzed (Participants) | 0 | 26 | 47
Participants | 0 | 23 | 35

2. Other Pre Specified Outcome: Patient Survival With Early Versus Standard of Care NIPPV Treatment
Description: Duration of patient survival
Time Frame: one year
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Compliance With NIPPV Treatment
Description: Number of hours of NIPPV use per month
Time Frame: one month
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Total Daily Energy Expediture (TDEE) of ALS Patients
Description: Total daily energy expenditure (TDEE) with be measured using the dual labeled water (DLW) method
Time Frame: Duration of study (approximately 1 year)
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Tolerance of NIPPV Treatment
Description: Percent of patients achieving tolerance (>4hr/night NIPPV after 2-3 week titration period) determined by actual usage data.
Time Frame: one month
Population: No data were collected for the "Standard of Care NIIPPV and Nutritional Monitoring" arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care NIPPV and Nutritional Monitoring | Standard of Care NIPPV | Early NIPPV
Number analyzed (Participants) | 0 | 23 | 35
Participants | 0 | 11 | 14

ADVERSE EVENTS:
Time Frame: 3 years, 4 months
Groups:
- Combined Arms: Sincere efforts were made to locate per arm data, but these data are no longer available. All adverse events are reported as one arm/group.
Arm/Group | Combined Arms
All-Cause Mortality (participants affected / at risk) | 19/153
Serious Adverse Events (participants affected / at risk) | 42/153
Other Adverse Events (participants affected / at risk) | 62/153
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined Arms (N=153)
ALS Progression (Nervous system disorders) | 1 (1) — Dates: 5/5/2007 5/25/2007 Status: Resolved Reason for Qualifying: Are other conditions which represent significant hazards Intensity: Moderate Relationship to study: Unrelated Description: Treatment and Evaluation of ALS Progression
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Dates: 5/11/2008 5/12/2008 Status: Resolved Reason for Qualifying: Requiring or prolonging hospitalization Intensity: Mild Relationship to study: Unrelated Description: Aspiration
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Dates: 6/10/2007 6/19/2007 Status: Resolved Reason for Qualifying: Requiring or prolonging hospitalization Intensity: Moderate Relationship to Study: Unrelated Description: Presumed Aspiration Pneumonia
Bladder malignancy/UTI (Renal and urinary disorders) | 1 (1) — Dates: 8/22/2007 9/5/2007 Status: Resolved Reason for qualifying: Requiring or prolonging hospitalization Intensity: Severe Relationship to Study: Unrelated Description: Possible bladder malignancy and UTI
Blood Clot (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Dates: 8/21/2005 9/1/2005 Status:Resolved Reason for Qualifying: Requiring or prolonging hospitalization Intensity: Moderate Relationship to study: Unrelated Description: Blood Clot Behind right knee
Cardiac Arrest (Cardiac disorders) | 1 (1) — Dates: 4/4/2006 4/4/2006 Status: Resolved Reason for Qualifying: Resulting in death Intensity: Severe Relationship to Study: Unrelated Description: Cardiac Arrest
Colonic Bleed (Gastrointestinal disorders) | 1 (1) — Dates: 1/15/2007 1/29/2007 Status: Resolved Reason for Qualifying: Requiring or prolonging hospitalization Intensity: Severe Relationship: Unrelated Description: Left Colonic Bleed
Concussion (Nervous system disorders) | 1 (1) — Dates: 2/7/2007 2/7/2007 Status: Resolved Reason for Qualifying: Life-threatening Intensity: Moderate Relationship to Study: Unrelated Description: Concussion as result of Automobile Accident
Death (General disorders) | 14 (14) — Dates: 6/2/2006 6/2/2006 Status: Resolved Reason for Qualifying: Resulting in death Intensity: Severe Relationship to Study: Unrelated Description: No Information Given
Difficulty Breathing (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Dates: 5/21/2007 5/27/2007 Status: Resolved Reason for Qualifying: Requiring or prolonging hospitalization Intensity: Moderate Relationship to Study: Unrelated Description: Difficulty breathing due to Sialorrhea
Dislodged PEG Tube (Gastrointestinal disorders) | 1 (1) — Dates: 6/30/2007 Status: Continuing at discontinuation Reason for Qualifying: Requiring or prolonging hospitalization Intensity: Severe Relationship to Study: Unrelated Description: Dislodged PEG Tube and Respiratory Distress
Distended Abdomen (Gastrointestinal disorders) | 1 (1) — Dates: 8/24/2005 8/29/2005 Status: Resolved Reason for Qualifying: Requiring or prolonging hospitalization Intensity: Moderate Relationship to Study: Unrelated Description: Distended Abdomen
Dysphagia (Gastrointestinal disorders) | 3 (3) — Dates: 3/11/2008 3/11/2008 Status: Resolved Reason for Qualifying: Requiring or prolonging hospitalization Intensity: Severe Relationship to study: Unrelated Description: Dysphagia
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Dates: 4/9/2007 Status: Continuing at discontinuation Reason for Qualifying: Requiring or prolonging hospitalization Intensity: Severe Relationship to study: Unrelated Description: Increased Dyspnea
Failure to Thrive (Metabolism and nutrition disorders) | 1 (1) — Dates: 7/23/2007 8/10/2007 Status: Resolved Reason for Qualifying: Requiring or prolonging hospitalization Intensity: Moderate Relationship to Study: Unrelated Description: Diagnosed as failure to thrive
Hip Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Dates: 4/25/2006 5/4/2006 Status: Resolved Reason for Qualifying: Requiring or prolonging hospitalization Intensity: Moderate Relationship to study: Unrelated Description: Left Hip Fracture Resulting From Fall
Hypokalemia, hypomagnesia, and antythmia (Metabolism and nutrition disorders) | 1 (1) — Dates: 12/15/2007 12/17/2007 Status: Resolved Reason for qualifying: Requiring or prolonging hospitalization Intensity: Severe Relationship to study: Unrelated Description: Hypokalemia, hypomagnesia, and antythmia
Infection (Infections and infestations) | 2 (2) — Dates: 10/3/2007 10/11/2007 Status: Resolved Reason for Qualifying: Requiring or prolonging hospitalization Intensity: Severe Relationship to study: Unrelated Description: Severe infection
Irregular Heartbeat (Cardiac disorders) | 2 (2) — Dates: 1/18/2008 2/17/2008 Status: Resolved Reason for Qualifying: Requiring or prolonging hospitalization Intensity: Severe Relationship to study: Unrelated Description: Irregular Heartbeat
Laceration (Skin and subcutaneous tissue disorders) | 1 (1) — Dates: 9/9/2007 11/4/2007 Status: Resolved Reason for Qualifying: Requiring or prolonging hospitalization Intensity: Severe Relationship to Study: Unrelated Description: Debridement and Closure of Laceration
Liver Cancer Diagnosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Dates: 11/4/2005 Status: Continuing at discontinuation Reason for Qualifying: Are other conditions which represent significant hazards Intensity: Severe Relationship to Study: Unrelated Description: Liver Cancer Diagnosis
Loculated right pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Dates: 7/27/2007 8/2/2007 Status: Resolved Reason for qualifying: Requiring or prolonging hospitalization Intensity: Severe Relationship to Study: Unrelated Description: Loculated right pleural effusion and possible Pneumonia
Myocardial Infarction (Cardiac disorders) | 1 (1) — Dates: 8/30/2007 8/31/2007 Status: Resolved Reason for Qualifying: Requiring or prolonging hospitalization Intensity: Severe Relationship to study: Unrelated Description: Apparent Myocardial Infarction
PEG Procedure Complications (Gastrointestinal disorders) | 2 (2) — Dates: 5/11/2006 5/12/2006 Status: Resolved Reason for Qualifying: Requiring or prolonging hospitalization Intensity: Moderate Relationship to study: Unrelated Description: Complications from PEG Procedure
Peg Replacement (Surgical and medical procedures) | 2 (2) — Dates: 3/14/2008 3/18/2008 Status: Resolved Reason for qualifying: Requiring or prolonging hospitalization Intensity: Mild Relationship to study: Unrelated Description: PEG replacement
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 4 (4) — Dates: 3/6/2008 3/19/2008 Status: Resolved Reason for qualifying: Requiring or prolonging hospitalization Intensity: Severe Relationship to study: Unrelated Description: Pneumonia
Pulmonary Emboli and pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Dates: 9/3/2006 10/5/2006 Status: Resolved Reason for Qualifying: Requiring or prolonging hospitalization Intensity: Severe Relationship to study: Unrelated Description: Pulmonary emboli and pneumonia
Respiratory Complications (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Dates: 10/7/2006 10/7/2006 Status: Resolved Reason for Qualifying: Resulting in death Intensity: Severe Relationship to study: Unrelated Description: Respiratory Complications
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Dates: 9/28/2007 9/28/2007 Status: Resolved Reason for qualifying: Requiring or prolonging Hospitalization Intensity: Severe Relationship to study: Unrelated Description: continued respiratory decline
Sepsis (Gastrointestinal disorders) | 1 (1) — Dates: 10/3/2007 10/11/2007 Status: Resolved Reason for Qualifying: Requiring or prolonging hospitalization Intensity: Severe Relationship to Study: Unrelated Description: Severe Sepsis around PEG Tube
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Dates: 10/2/2006 Status: Continuing at discontinuation Reason for Qualifying: Are other conditions which represent significant hazards Intensity: Severe Relationship: Unrelated Description: Shortness of breath
Subarachroid Hemmorrhage and Contusion (Skin and subcutaneous tissue disorders) | 1 (1) — Dates: 3/14/2007 3/16/2007 Status: Resolved Reason for Qualifying: Resulting in death Severe Relationship to Study: Unrelated Description: Sub-arachnoid Haemmorrhage and Contusion Resulting from fall
Subdural Hematoma (Skin and subcutaneous tissue disorders) | 1 (1) — Dates: 6/11/2007 6/11/2007 Status: Resolved Reason for Qualifying: Requiring or prolonging hospitalization Intensity: Severe Relationship to Study: Unrelated Description: Subdural Hematoma from fall
Transitional Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Dates: 9/6/2007 9/23/2007 Status: Resolved Reason for Qualifying: Resulting in death Intensity: Severe Relationship to study: Unrelated Description Small bowel obstruction, transitional cell carcinoma
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combined Arms (N=153)
Abdominal Distension (Gastrointestinal disorders) | 3 (3) — Dates: 3/20/2007 Status: Unresolved at 48 Weeks Description: Abdominal distension Intensity: moderate Relationship to study: possible
Abnormal Lab (Metabolism and nutrition disorders) | 8 (8) — Dates: 5/2/2006 8/21/2006 Status: Resolved Description: Abnormal Lab Intensity: mild Relationship to study: not related
Allergy (Immune system disorders) | 2 (2) — Dates: 4/17/2007 4/22/2007 Status: Ended Description: Allergy Intensity: mild Relationship to study: not related
Ankle Sprain (Musculoskeletal and connective tissue disorders) | 1 (1) — Dates: 9/6/2006 Status: Ended Description: Ankle Sprain Intensity: moderate Relationship to study: not related
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) — Dates: 3/27/2007 Status: Unresolved at 48 Weeks Description: Arthritis Intensity: mild Relationship to study: not related
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4) — Dates:: 6/3/2006 Status: Unresolved at 48 weeks Description: Back Pain Intensity: moderate Relationship to study: not related
Blister (Skin and subcutaneous tissue disorders) | 1 (1) — Dates: 4/1/2008 Status: Unresolved at 48 Weeks Description: Blister Intensity: mild Relationship to study: not related
Blood Clot (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Dates: 1/28/2008 Status: Unresolved at 48 Weeks Description: Blood Clot Intensity: moderate Relationship to study: not related
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) — Dates: 1/20/2008 2/10/2008 Status: Ended Description: Bronchitis Intensity: moderate Relationship to study: possible
Bruise (Skin and subcutaneous tissue disorders) | 2 (2) — Dates: 5/11/2006 5/11/2006 Status:Ended Description: Bruise Intensity: mild Relationship to study: not related
Burning Sensation (General disorders) | 1 (1) — Dates: 7/23/2007 Status: Continuing Description: PAIN Burning Sensation Intensity: severe Relationship to study: not related
Cold (General disorders) | 7 (8) — Dates: 8/9/2007 8/15/2007 Status: Ended Description: Cold Intensity: mild Relationship to study: not related
Colon Polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Dates: 2/1/2006 2/1/2006 Status: Ended Description: Colon Polyp Intensity: mild Relationship: not related
Concussion (Nervous system disorders) | 1 (1) — Dates: 2/6/2006 2/6/2006 Status: Ended Description: Concussion Intensity: severe Relationship to study: not related
Congestion (Immune system disorders) | 2 (2) — Dates: 7/21/2006 7/31/2006 Status: Resolved Description: Congestion Intensity: moderate Relationship to study: not related
Conjunctivitis (Infections and infestations) | 2 (2) — Dates: 7/3/2007 7/8/2007 Status: Ended Description: Conjunctivitis Intensity: mild Relationship to study: not related
Constipation (Gastrointestinal disorders) | 8 (8) — Dates: 2/1/2006 6/1/2006 Status: Resolved Description: Constipation Intensity: moderate Relationship to study: not likely
Contusion (Skin and subcutaneous tissue disorders) | 1 (1) — Dates: 7/4/2007 7/4/2007 Status: Ended Description: Contusion Intensity: mild Relationship to study: not related
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Dates: 9/7/2006 Status: Ended Description: Cough Intensity: moderate Relationship: not related
Decreased Rectal Tone (Gastrointestinal disorders) | 1 (1) — Dates: 6/4/2007 Status: Continuing Description: Decreased Rectal Tone Intensity: moderate Relationship to study: not related
Dehydration (Gastrointestinal disorders) | 1 (1) — Dates: 3/5/2008 Description: Dehydration Intensity: mild Relationship to study: not likely
Dental (Gastrointestinal disorders) | 1 (1) — Dates: 4/17/2006 Status: Ended Description: Dental Intensity: moderate Relationship to study: not related
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) — Dates: 3/1/2008 Status: Unresolved at 48 Weeks Description: Dermatitis Intensity: mild Relationship to study: possible
Diarrhea (Gastrointestinal disorders) | 4 (6) — Dates: 2/10/2007 2/10/2007 Status: Ended Description: Diarrhea Intensity: mild Relationship to study: not related
Diverticulitis (Gastrointestinal disorders) | 1 (1) — Dates: 10/15/2006 11/14/2006 Status: Resolved Description: Diverticulitis Intensity: severe Relationship to study: not related
Dizziness (Nervous system disorders) | 3 (4) — Dates: 1/15/2006 Status: Ended Description: Dizziness Intensity: moderate Relationship to study: not related
Dry Eye (Eye disorders) | 1 (1) — Dates: 10/15/2007 Description:Dry Eye Intensity: mild Relationship to study: probable
Dysphagia (Gastrointestinal disorders) | 1 (1) — Dates: 6/15/2006 Status: Unresolved at 48 Weeks Description: Dysphagia Intensity: mild Relationship to study: not likely
Ear Infection (Infections and infestations) | 1 (1) — Dates: 10/1/2006 10/26/2006 Status: Resolved Description: Ear Infection Intensity: mild Relationship to study: not related
Edema (Blood and lymphatic system disorders) | 7 (7) — Dates: 10/24/2006 Status: Unresolved at 48 Weeks Description: Edema Intensity: mild Relationship to study: not likely
Fall (General disorders) | 8 (9) — Dates: 4/13/2007 4/13/2007 Status: Ended Description: Fall Intensity: mild Relationship to study: not related
Fatigue (General disorders) | 5 (5) — Dates: 11/1/2005 Status: Unresolved at Discontinuation Description: Fatigue Intensity: severe Relationship to study: not related
Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Dates: 1/18/2007 3/29/2007 Status: Resolved Description: Fracture Intensity: mild Relationship to study: not related
Gastritis (Gastrointestinal disorders) | 1 (1) — Dates: 9/25/2006 10/2/2006 Status: Ended Description: Gastritis Intensity: severe Relationship to study: not related
Hallucination (Nervous system disorders) | 1 (1) — Dates: 9/13/2006 9/16/2006 Status: Ended Description: Hallucination Intensity: moderate Relationship to study: not related
Headache (Nervous system disorders) | 2 (2) — Dates: 1/18/2006 3/1/2006 Status: Ended Description: Headache Intensity: mild Relationship to study: not related
Hypercarbia (Metabolism and nutrition disorders) | 1 (1) — Dates: 11/6/2006 Status: Continuing Description: Hypercarbia Intensity: mild Relationship to study: not related
Hypertension (Cardiac disorders) | 1 (1) — Dates: 1/11/2008 Status: Unresolved at 48 Weeks Description: Hypertension Intensity: mild Relationship to study: not likely
Hypotension (Cardiac disorders) | 1 (1) — Dates: 11/4/2006 11/4/2006 Status: Ended Description: Hypotension Intensity: mild Relationship to Study: not related
Infection (Infections and infestations) | 1 (1) — Dates: 10/26/2007 11/4/2007 Status: Ended Description: Infection Intensity: mild Relationship to study: not related
Knee Sprain (Musculoskeletal and connective tissue disorders) | 1 (1) — Dates: 6/30/2007 7/13/2007 Status: Ended Description: Knee Sprain Intensity: moderate Relationship to study: not related
Laceration (Skin and subcutaneous tissue disorders) | 2 (3) — Dates: 2/5/2007 2/5/2007 Status: Ended Description: Laceration Intensity: mild Relationship to study: not related
Lesion (Skin and subcutaneous tissue disorders) | 1 (1) — Dates: 3/30/2007 5/7/2007 Status: Ended Description: Lesion Intensity: mild Relationship to study: definite
Nosebleed (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Dates: 11/1/2007 Status: Continuing Description: Nosebleed Intensity: mild Relationship to study: probable
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) — Dates: 9/4/2006 Status: Unresolved at 48 Weeks Description: Osteopenia Intensity: mild Relationship to study: not likely
PEG (Gastrointestinal disorders) | 3 (3) — Dates: 6/29/2006 7/1/2006 Status: Ended Description: PEG Intensity: moderate Relationship to study: not related
Pain (General disorders) | 4 (6) — Dates: 11/20/2006 12/18/2006 Status: Resolved Description: Pain Intensity: moderate Relationship to study: not related
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Dates: 11/1/2007 Status: Unresolved at 48 Weeks Description: Pneumonia Intensity: moderate Relationship to study: not related
Post Nasal Drip (Immune system disorders) | 2 (2) — Dates: 3/31/2006 Status: Unresolved at 48 Weeks Description: Post Nasal Drip Intensity: severe Relationship to study: not related
Pressure Sores (Skin and subcutaneous tissue disorders) | 1 (2) — Dates: 11/28/2006 11/30/2006 Status: Resolved Description: Pressure Sores Intensity: mild Relationship to study: not related
RADS (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Dates: 1/17/2007 4/30/2007 Status: Ended Description: RADS Intensity: mild Relationship: not related
Rash (Skin and subcutaneous tissue disorders) | 4 (4) — Dates: 8/15/2005 Status: Unresolved at 48 Weeks Description: Rash Intensity: mild Relationship to study: not likely
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Dates: 2/25/2007 2/25/2007 Status: Ended Description: Shortness of Breath Intensity: moderate Relationship to study: not related
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 3 (3) — Dates: 1/23/2006 1/25/2006 Status: Ended Description: Shoulder Pain Intensity: severe Relationship to study: not related
Sialorrhea (Gastrointestinal disorders) | 1 (3) — Dates: 2/10/2006 Status: Unresolved at 48 Weeks Description: Sialorrhea Intensity: mild Relationship to study: not related
Sinus Infection (Infections and infestations) | 1 (1) — Dates: 4/1/2007 4/7/2007 Status: Ended Description: Sinus Infection Severity: moderate Relationship to study: not related
Sore Throat (General disorders) | 1 (2) — Dates: 10/12/2006 Status: Unresolved at 48 Weeks Description: Sore Throat Intensity: mild Relationship to study: not related
Spasm (Respiratory) (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Dates: 1/19/2007 1/19/2007 Status: Resolved Description: Spasm Intensity: mild Relationship to study: not related
Stomach Upset (Gastrointestinal disorders) | 3 (3) — Dates: 4/29/2006 5/1/2006 Status: Ended Description: Stomach Upset Intensity: mild Relationship to study: not related
UTI (Infections and infestations) | 4 (5) — Dates: 3/14/2006 3/24/2006 Status: Ended Description: UTI Intensity: moderate Relationship to study: not related
Urgent Bowel Movements (Gastrointestinal disorders) | 1 (1) — Dates: 2/1/2006 Status: Unresolved at Discontinuation Description: Urgent Bowel Movements Intensity: mild Relationship to study: possible
Urinary Frequency (Renal and urinary disorders) | 1 (1) — Dates: 6/11/2007 6/24/2007 Status: Ended Description: Urinary Frequency Intensity: moderate Relationship to study: not likely
Vomiting (Gastrointestinal disorders) | 1 (1) — Dates: 10/18/2005 10/18/2005 Status: Ended Description: Vomiting Intensity: mild Relationship to study: not related
Weakness (Musculoskeletal and connective tissue disorders) | 3 (4) — Dates: 2/1/2006 Status: Unresolved at Discontinuation Description: Weakness Intensity: mild Relationship to study: not related
Weight Loss (General disorders) | 1 (1) — Dates: 8/8/2005 3/13/2006 Status: Ended Description: Weight Loss Intensity: moderate Relationship to study: not related
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Dates: 11/6/2006 Status: Resolved Description: Wheezing Intensity: moderate Relationship to study: not related

LIMITATIONS AND CAVEATS:
Compliance with NIPPV intervention is limited due to technical difficulties in obtaining BiPAP download data from some sites. This was due to variability in the local respiratory therapists engaged by commercial respiratory therapy companies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes